CLINICAL TRIAL: NCT04606407
Title: Prospective, Open-label, Randomized, Multi-Center Study for Safety and Efficacy Evaluation of Inhaled Nitric Oxide (NO) Given Intermittently to Adults With Viral Pneumonia
Brief Title: Inhaled NO for the Treatment of Viral Pneumonia in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beyond Air Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA_VPLF_01
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Viral Pneumonia; Nitric Oxide; Respiratory Disease; Pneumonia, Viral; Inhaled Nitric Oxide; Covid19; SARS-CoV Infection
Keywords: Inhaled Nitric Oxide; iNO; Virus; Respiratory Disease; Viral Pneumonia; COVID-19; SARS-CoV-2
MeSH Terms: conditions — Pneumonia, Viral; Respiration Disorders; COVID-19; Severe Acute Respiratory Syndrome; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Treatment (Experimental): Inhaled NO delivered using LungFit™ in addition to standard of care
  Interventions: Device: LungFit™
- Standard of care (No Intervention): Standard of care

INTERVENTIONS:
Device: LungFit™ — Patients will receive inhalations of 150 ppm for 40 min 4 times a day, up to 7 days (maximum 28 treatments)
  Arms: Treatment

SUMMARY:
The purpose of this multi center, open label, randomized, study is to obtain information on the safety and efficacy of 150 ppm Nitric Oxide given in addition to the standard of care of patients with viral pneumonia

ELIGIBILITY:
Inclusion Criteria:

* Patients (male and female) admitted to the hospital for clinical diagnosis of viral pneumonia including COVID-19 patients that have a positive nasal swab.
* Age 18 to 80 years
* Female subjects must be willing to use medically acceptable contraception from screening to Day 30 (acceptable forms of contraception: abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent).
* Ability to understand and comply with study requirements.
* Signed informed consent by subject

Exclusion Criteria:

* Patients with pneumonia with two or more of the following:

  1. WBC of more than 15,000
  2. Lobar pneumonia
  3. Pleural effusion
* Patients who are treated with or require high flow nasal cannula, CPAP, intubation, mechanical ventilation, or tracheostomy
* Breastfeeding or pregnancy as evidenced by a positive pregnancy test.
* Subjects diagnosed with immunodeficiency, with history of congestive or unstable heart disease, left ventricular dysfunction (LVEF <40%) or myocardial damage, severe pulmonary hypertension and/or unstable hypertension
* Use of an investigational drug during the last 30 days prior enrollment
* Methemoglobin level >3% at screening
* Patients on chronic (over two weeks of treatment) systemic steroids (any formulation, excluding Dexamethasone or Prednisone) within 30 days prior to enrollment.
* History of daily, continuous oxygen supplementation
* Patients with BMI greater than or equal to 40
* Patients with clinically significant anemia, e.g., Hb <10.0 and/or thrombocytopenia, e.g., Platelets <75.
* Smokers who are unwilling to refrain from smoking during hospitalization
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data, e.g., known or suspected thalassemia, sickle cell disease or other diseases associated with poor oxygen carrying capacity.
* The subject is identified by the investigator as being unable or unwilling to perform study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-08-07 (Actual); Study Completion 2022-08-07 (Actual)

PRIMARY OUTCOMES:
incidence of Serious Adverse Events | 30 days
  Clinical safety will be assessed by incidence of Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
fever resolution | Baseline to 30 days
  Time to fever resolution
ICU admission | Baseline to 30 days
  Number of patients requiring admission to ICU
Oxygen support | Baseline to 30 days
  Time until patient no longer requires supportive oxygen
Stable room air saturation | Baseline to 30 days
  b.d. Stable room air saturation of 93% and above or returning to baseline saturation, whichever is lower

CONTACTS AND LOCATIONS:
Overall Officials: Asher Tal, Study Director — Beyond Air
Locations (3):
- Israel (3):
  - Shaare Zedek Medical Center, Jerusalem
  - Hasharon Medical Center, Petah Tikva
  - Rabin Medical Center, Petah Tikva

IPD SHARING:
Plan to Share IPD: No